CLINICAL TRIAL: NCT01506856
Title: A Randomized Phase II/III Trial of Intravenous (IV) Paclitaxel Weekly Plus IV Carboplatin Once Every 3 Weeks Versus IV Paclitaxel Weekly Plus Intraperitoneal (IP) Carboplatin Once Every 3 Weeks in Women With Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Intraperitoneal Therapy For Ovarian Cancer With Carboplatin Trial
Acronym: iPocc
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Trial & Investigation Consortium (Network)
Collaborators: Japanese Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOTIC-001/JGOG3019; UMIN000003670 (Other Grant/Funding Number: University Hospital Medical Information Network = UMIN); jRCTs031180141 (Other Grant/Funding Number: jRCT（Japan Registry of Clinical Trials）)
Record Dates: First submitted 2011-12-20; First posted 2012-01-10 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2022-09

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Epithelial ovarian cancer; Fallopian tube cancer; peritoneal cancer; intraperitoneal therapy; Carboplatin; Paclitaxel
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment: dd-TCiv therapy (Active Comparator): Paclitaxel administered by IV infusion weekly plus concurrent carboplatin administered by IV infusion once every 3 weeks
  Interventions: Drug: Paclitaxel(intravenous) + Carboplatin(intravenous)
- Study treatment: dd-TCip therapy (Experimental): Paclitaxel administered by IV infusion weekly plus concurrent carboplatin administered by IP injection once every 3 weeks
  Interventions: Drug: Paclitaxel(intravenous) + Carboplatin(intraperitoneal)

INTERVENTIONS:
Drug: Paclitaxel(intravenous) + Carboplatin(intravenous) — Paclitaxel(intravenous) + Carboplatin(intravenous) Paclitaxel : 80mg/m2, IV infusion, Day1, 8, and 15 Carboplatin: AUC=6.0, IV infusion, Day1 A total of 6 to 8 cycles will be repeated.
  Other Names: Paclitaxel(Sawai),(NK), Paraplatin(BMS), Carboplatin(SANDOZ)
  Arms: Standard treatment: dd-TCiv therapy
Drug: Paclitaxel(intravenous) + Carboplatin(intraperitoneal) — Paclitaxel(intravenous) + Carboplatin(intraperitoneal) Paclitaxel : 80mg/m2, IV infusion, Day1, 8, and 15 Carboplatin: AUC=6.0, IP injection, Day1 A total of 6 to 8 cycles will be repeated.
  Other Names: Paclitaxel(Sawai),(NK), Paraplatin(BMS), Carboplatin(SANDOZ)
  Arms: Study treatment: dd-TCip therapy

SUMMARY:
The purpose of this study is:

Phase A: To confirm the feasibility of paclitaxel administered by intravenous (IV) infusion weekly plus concurrent carboplatin administered by intraperitoneal (IP) injection once every 3 weeks (dd-TCip therapy).

Phase B: To compare the efficacy and safety of the following two treatment regimens as first-line chemotherapy in women with epithelial ovarian, Fallopian tube or primary peritoneal cancer.

DETAILED DESCRIPTION:
This is a randomized, multicenter international study. Patient are stratified according to Residual tumor diameter([0cm(No residual)] vs. [0cm<residual<1cm] vs. [1cm<residual<2cm] vs. [>2 cm]), FIGO stage(StageII vs. III vs. IV) and institution. Patient randomized to one of the treatment arms described below.

RegimenI(Standard treatment: dd-TCiv therapy): Paclitaxel administered by IV infusion weekly plus concurrent carboplatin administered by IV infusion once every 3 weeks

RegimenII(Study treatment: dd-TCip therapy): Paclitaxel administered by IV infusion weekly plus concurrent carboplatin administered by IP injection once every 3 weeks

The 3-week period (21 days) is 1 cycle. Protocol treatment basically comprises 6 cycles. IDS is allowed to be performed after 3, 4 or 5 cycles of the protocol treatment. In such cases, the protocol treatment must be restarted within 8 weeks after IDS. If IDS is performed, patients can receive up to 3 additional cycles of the protocol treatment after IDS. If interval debulking surgery (IDS) is performed after 3, 4 or 5 cycles, the patients can receive up to 3 additional cycles of the protocol treatment. A total of 6 to 8 cycles will be repeated.

The analysis of efficacy will be performed on all randomized subjects in accordance with the intention-to-treat (ITT) principle. In order to assess the robustness of the results, the same analyses will be done using all randomized subjects who satisfy the eligibility criteria. The analysis of safety will be performed on all subjects who have received at least one dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients assumed to have a stageII-IV epithelial ovarian, fallopian tube, or primary peritoneal cancer as a pre-surgery diagnosis
2. Patients scheduled to undergo laparotomy

   *Both optimal and suboptimal patients will be eligible for the study (Suboptimal patients, as well as those who undergo only exploratory laparotomy, are eligible.)
3. ECOG Performance Status: 0-2
4. Patients who provide consent for placement of the IP port system, if randomized to Regimen II (Study treatment: dd-TCip therapy)
5. Patients expected to receive the first protocol treatment within 8 weeks after the comprehensive staging surgery
6. Lab data and clinical examination: Data within 28 days before the scheduled date of surgery

   * Neutrophil count ≧ 1,500 /mm3
   * Platelet count ≧ 100,000 /mm3
   * AST (GOT) ≦ 100 IU/L
   * ALT (GPT) ≦ 100 IU/L
   * Total bilirubin < 1.5 mg/dL
   * Serum Creatinine < 1.5 mg/dL
   * Electrocardiogram (ECG): Patients with normal ECG, Asymptomatic patients with abnormal ECGs not requiring medical intervention
   * Neuropathy(Both motor and sensory) ≦ Grade1 (CTCAE Version 4.0)
7. Patients expected to survive longer than 3 months from the start date of the protocol treatment
8. Patients aged 20 years and older at the time of tentative registration (with no upper age limit)
9. Patients who provide written informed consent for participation in this trial

Exclusion Criteria:

1. Patients assumed to have a borderline malignancy of the ovary, fallopian tube, or primary peritoneal cancer
2. Patients who have received previous chemotherapy or radiation therapy to treat the current disease
3. Patients who have a synchronous malignancy or who have been progression-free less than 5 years for a metachronous malignancy (Patients with basal and squamous cell carcinoma of the skin, as well as carcinoma in situ, and intramucosal carcinoma cured by local treatment, are eligible for the study)
4. Patients with serious medical complications, such as serious heart disease, cerebrovascular accidents, uncontrolled diabetes mellitus, uncontrolled hypertension, pulmonary fibrosis, interstitial pneumonitis, active bleeding, an active gastrointestinal ulcer, or a serious neurological disorder
5. Patients who have had a hypersensitivity reaction to polyoxyethylated or hydrogenated castor oil
6. Patients with a pleural effusion requiring continuous drainage
7. Patients with an active infection requiring antibiotics
8. Patients who are pregnant, nursing or of child-bearing potential
9. Patients with evidence upon physical examination of brain tumor and any brain metastases
10. Patients for whom completion of this study and/or follow-up is deemed inappropriate for any reason
11. Patients with any signs/symptoms of interstitial pneumonia

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2010-05; Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed until 510 events are observed or until 3 years from the last patient is randomized to the study

SECONDARY OUTCOMES:
Overall survival (OS) | weekly during the protocl treatment, then every 3 months for the first 2 years, 6-month for the following 2 years, and once a year thereafter
Tumor response (only patients with evaluable disease) | every 2 cycles [after 2 cycles, after 4 cycles, after 6 cycles, (after 8 cycles)], the time of discontinuation of the protocol treatment and then at least annually during follow-up
Adverse events | weekly during the protocl treatment, then every 3 months for the first 2 years, 6-month for the following 2 years, and once a year thereafter
Treatment completion rate | After the last cycle of the protocol teatment
Quality of Life (QOL) assessments | baseline, after 3 cycles, 6 cycles, 36 week, 60 weeks and 84 weeks from the start of protocol treatment
Cost-utility analysis | baseline, after 3 cycles, 6 cycles, 36 week, 60 weeks and 84 weeks from the start of protocol treatment

CONTACTS AND LOCATIONS:
Overall Officials: Keiichi Fujiwara, MD, PhD, Study Chair — Saitama Medical University International Medical Center Comprehensive Cancer Center
Locations (62):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States
- Queen Mary Hospital, Hong Kong, High West, Hong Kong
- Japan (52):
  - Aichi Cancer Center Hospital, Chikusa, Aichi-ken
  - Hirosaki University School of Medicine & Hospital, Hirosaki-shi, Aomori
  - The Jikei University School of Medicine, Kashiwa Hospital, Kashiwa, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Toon-shi, Ehime
  - University of Fukui Hospital, Yoshida, Fukui
  - Gunma University Hospital, Maebashi, Gunma
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - NHO Kure Medical Center And Chugoku Cancer Center, Kure, Hiroshima
  - Miyoshi Central Hospital, Miyoshi, Hiroshima
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Japanese Red Cross Society Himeji Hospital, Himeji, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Hyogo Medical College Hospital, Nishinomiya, Hyōgo
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Nippon Medical University Musasi Kosugi Hospital, Kawasaki-shi, Kanagawa
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Mie Prefectural General Medical Center, Yokkaichi, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto, Nagano
  - Nara Medical Univeｒsity Hospital, Kashihara, Nara
  - Okinawa Prefectural Chubu Hospital, Uruma, Okinawa
  - Kaizuka City Hospital, Kaizuka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Saitama Medical University Saitama Medical Center, Kawagoe, Saitama
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Juntendo University Hospital, Bunkyo, Tokyo
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - The Jikei University Daisan Hospital, Komae, Tokyo
  - The Cancer Institute Hospital Of JFCR, Koto-Ku, Tokyo
  - The Jikei University Hospital, Minato-Ku, Tokyo
  - Showa University Hospital, Shinagawa-Ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Tokyo Women's Medical University Medical Center East, Shinjuku-Ku, Tokyo
  - Tottori University, Yonago, Tottori
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - NHO Kyusyu Medical center, Fukuoka
  - JA Hiroshima General Hospital, Hiroshima
  - Kagoshima City Hospital, Kagoshima
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Saiseikai Nagasaki Hospital, Nagasaki
  - Niigata Cancer Center Hospital, Niigata
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Tottori Municipal Hospital, Tottori
- University of Otago - Christchurch/Christchurch Women's Hospital, Christchurch, New Zealand
- Singapore (2):
  - KK Women's and Children's Hospital, Bukit Timah
  - National University Hospital of Singapore, Kent Ridge
- South Korea (5):
  - Korea Cancer Center Hospital, Seoul, Gongneung-Dong
  - Gangnam Severance Hospital in Korea, Dogok, Seoul
  - Asan Medical Center, P’ungnap-tong, Seoul
  - Ewha Womans University Medical Center, Yangcheon, Seoul
  - Shinchon Severance Hospital, Seoul, Shinchon

REFERENCES:
- [Background] Bristow RE, Tomacruz RS, Armstrong DK, Trimble EL, Montz FJ. Survival effect of maximal cytoreductive surgery for advanced ovarian carcinoma during the platinum era: a meta-analysis. J Clin Oncol. 2002 Mar 1;20(5):1248-59. doi: 10.1200/JCO.2002.20.5.1248. PMID 11870167
- [Background] Neijt JP, Engelholm SA, Tuxen MK, Sorensen PG, Hansen M, Sessa C, de Swart CA, Hirsch FR, Lund B, van Houwelingen HC. Exploratory phase III study of paclitaxel and cisplatin versus paclitaxel and carboplatin in advanced ovarian cancer. J Clin Oncol. 2000 Sep;18(17):3084-92. doi: 10.1200/JCO.2000.18.17.3084. PMID 10963636
- [Background] Piccart MJ, Bertelsen K, James K, Cassidy J, Mangioni C, Simonsen E, Stuart G, Kaye S, Vergote I, Blom R, Grimshaw R, Atkinson RJ, Swenerton KD, Trope C, Nardi M, Kaern J, Tumolo S, Timmers P, Roy JA, Lhoas F, Lindvall B, Bacon M, Birt A, Andersen JE, Zee B, Paul J, Baron B, Pecorelli S. Randomized intergroup trial of cisplatin-paclitaxel versus cisplatin-cyclophosphamide in women with advanced epithelial ovarian cancer: three-year results. J Natl Cancer Inst. 2000 May 3;92(9):699-708. doi: 10.1093/jnci/92.9.699. PMID 10793106
- [Background] Ozols RF, Bundy BN, Greer BE, Fowler JM, Clarke-Pearson D, Burger RA, Mannel RS, DeGeest K, Hartenbach EM, Baergen R; Gynecologic Oncology Group. Phase III trial of carboplatin and paclitaxel compared with cisplatin and paclitaxel in patients with optimally resected stage III ovarian cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2003 Sep 1;21(17):3194-200. doi: 10.1200/JCO.2003.02.153. Epub 2003 Jul 14. PMID 12860964
- [Background] Katsumata N, Yasuda M, Takahashi F, Isonishi S, Jobo T, Aoki D, Tsuda H, Sugiyama T, Kodama S, Kimura E, Ochiai K, Noda K; Japanese Gynecologic Oncology Group. Dose-dense paclitaxel once a week in combination with carboplatin every 3 weeks for advanced ovarian cancer: a phase 3, open-label, randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1331-8. doi: 10.1016/S0140-6736(09)61157-0. Epub 2009 Sep 18. PMID 19767092
- [Background] Alberts DS, Liu PY, Hannigan EV, O'Toole R, Williams SD, Young JA, Franklin EW, Clarke-Pearson DL, Malviya VK, DuBeshter B. Intraperitoneal cisplatin plus intravenous cyclophosphamide versus intravenous cisplatin plus intravenous cyclophosphamide for stage III ovarian cancer. N Engl J Med. 1996 Dec 26;335(26):1950-5. doi: 10.1056/NEJM199612263352603. PMID 8960474
- [Background] Markman M, Bundy BN, Alberts DS, Fowler JM, Clark-Pearson DL, Carson LF, Wadler S, Sickel J. Phase III trial of standard-dose intravenous cisplatin plus paclitaxel versus moderately high-dose carboplatin followed by intravenous paclitaxel and intraperitoneal cisplatin in small-volume stage III ovarian carcinoma: an intergroup study of the Gynecologic Oncology Group, Southwestern Oncology Group, and Eastern Cooperative Oncology Group. J Clin Oncol. 2001 Feb 15;19(4):1001-7. doi: 10.1200/JCO.2001.19.4.1001. PMID 11181662
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] Miyagi Y, Fujiwara K, Kigawa J, Itamochi H, Nagao S, Aotani E, Terakawa N, Kohno I; Sankai Gynecology Study Group (SGSG). Intraperitoneal carboplatin infusion may be a pharmacologically more reasonable route than intravenous administration as a systemic chemotherapy. A comparative pharmacokinetic analysis of platinum using a new mathematical model after intraperitoneal vs. intravenous infusion of carboplatin--a Sankai Gynecology Study Group (SGSG) study. Gynecol Oncol. 2005 Dec;99(3):591-6. doi: 10.1016/j.ygyno.2005.06.055. Epub 2005 Aug 10. PMID 16095677
- [Background] Fujiwara K, Armstrong D, Morgan M, Markman M. Principles and practice of intraperitoneal chemotherapy for ovarian cancer. Int J Gynecol Cancer. 2007 Jan-Feb;17(1):1-20. doi: 10.1111/j.1525-1438.2007.00809.x. PMID 17291226
- [Background] Demets DL. Futility approaches to interim monitoring by data monitoring committees. Clin Trials. 2006;3(6):522-9. doi: 10.1177/1740774506073115. PMID 17170036
- [Background] Huang HQ, Brady MF, Cella D, Fleming G. Validation and reduction of FACT/GOG-Ntx subscale for platinum/paclitaxel-induced neurologic symptoms: a gynecologic oncology group study. Int J Gynecol Cancer. 2007 Mar-Apr;17(2):387-93. doi: 10.1111/j.1525-1438.2007.00794.x. PMID 17362317
- [Background] Calvert AH, Newell DR, Gumbrell LA, O'Reilly S, Burnell M, Boxall FE, Siddik ZH, Judson IR, Gore ME, Wiltshaw E. Carboplatin dosage: prospective evaluation of a simple formula based on renal function. J Clin Oncol. 1989 Nov;7(11):1748-56. doi: 10.1200/JCO.1989.7.11.1748. PMID 2681557
- See also: Japanese Gynecologic Oncology Group — http://www.jgog.gr.jp/